

Subject Informed Consent Form

Dubé A<sup>1</sup>., Brun C<sup>1</sup>., Albert WJ<sup>2</sup>. & Cardoso MR<sup>1</sup>.

Université de Moncton University of New Brunswick

June 7<sup>th</sup>, 2024

# **Subject Informed Consent Form**

## **CONSENT**

| The purpose of this study has been explained to me by I have understood the information, including the risks of participation, and agree to participate in the study. I have been given a copy of the Study Information sheet and the Consent form, which I have read and understood. I have been given an opportunity to ask questions about the study and my participation, and I understand that I may withdraw at any time. This project has been reviewed by the Research Ethics board of the University of New Brunswick and is on file as REB 2024-040 | | |
|---|---|---|
| during a manual material hand | participate in the study to be obse<br>ling task using a technique of my o<br>raw from it at any time, without pe | own selection, with the |
| Name of Participant (Print) | Signature of Participant | Date |
| Witness (Print) | Signature of Witness | Date |
| If you wish to be informed of the | e research results, please provide | contact information. |
| Name:<br>Telephone #:<br>Email address: | | |
| The researchers' contact infor Alexis Dubé, ead7300@umonct | <u>on.ca</u> , (506) 863-4342 | |
| Dr. Wayne Albert, walbert@unk | .cardoso@umoncton.ca, (506) 86. | 3-2033 |
| Other contact information: | | |

 $Assistant\ Dean-Graduate\ Studies:\ Jonathon\ Edwards,\ Jonathon.edwards@unb.ca$ 

#### **Letter of Information**

# An investigation of the physical task demands of caregivers working in a long-term care facility

### **Principal Investigators**

| Alexis Dubé, Student, bachelor's degree in Kinesiology<br>University de Moncton ead7300@umoncton.ca<br>(506) 864-4342 | Dr. Michelle Cardoso; Assistant Professor École de kinésiologie et de loisir, Université de Moncton Michelle.cardoso@umoncton.ca (506) 863-2033 |
|---|---|
| Dr. Wayne Albert Dean - Faculty of Kinesiology University of New Brunswick walbert@unb.ca, (506) 447-3254 | Chair of the UNB Research Ethics<br>Board:<br>Dr. David Coleman<br>ethics@unb.ca<br>(506) 453-5189 |

#### BACKGROUND AND PUROPOSE OF THIS STUDY

Healthcare workers, particularly caregivers in long-term care facilities, constitute a population at high risk of musculoskeletal injuries (MSIs) development at work (Gideon Asuquo et al., 2021). In Canada, the health care and social assistance sector accounted for more than 24% of total lost-time claims in 2021 (Statistics | AWCBC / ACATC, 2021). Musculoskeletal injuries account for over 83% of lost-time claims among healthcare professionals (Ngan et al., 2010). Work related musculoskeletal injuries are more prevalent among caregivers working in long-term care facilities compared to other nursing sectors, leading to over 63% leaving the profession for this reason (Gideon Asuquo et al., 2021).

The purpose of this study is to identify the physical tasks and demands of caregivers working in a long-term care facility. The results derived from this study will enable our research group to formulate a variety of strategies and intervention plans aimed at reducing the occurrence of work-related musculoskeletal injuries among caregivers. Solutions will vary; technological advancements, warm-up and stretching programs are examples of interventions that could potentially be beneficial for reducing the risks of injuries in the workplace.

#### WHAT WE ASK OF YOU:

#### TASK ANALYSIS TYPE OF STUDY

The study involves a researcher following you throughout your workday to quantify the physical tasks and demands of your occupation. If you choose to take part in this study, your workday will not be interrupted. It's important to note that the researchers present during the intervention are <u>not there to evaluate your job performance</u>, but rather to record the number of times each physical tasks and demands are performed throughout your shift. The time spent on different specific tasks will also be noted, as well as the number and duration of breaks during your working day. <u>These results will not be shared with your superiors</u>. The data we acquire will provide a more comprehensive insight into a typical workday in your field, enhancing our understanding of the factors contributing to the high rate of work-related injuries in this profession. At any time, if you or the residents are concerned about the presence of a researcher, you can mention it, and the researcher will leave you to take care of the resident alone.

Two pieces of non-invasive equipment will be used during data collection such as an Empatica (wristwatch) and a heart rate monitor (chest strap) to assess stress levels during your workday.

To monitor the level of perceived discomfort throughout the day, you will be asked to complete the Rate of Perceived Discomfort Questionnaire (RPD-Q) three times during your workday; specifically at the beginning, middle and at the end of your shift.

Additionally, The Health and Lifestyle questionnaire will be administered during data collection. Questions will cover your current levels of physical activity, sleeping patterns, general lifestyle, and any previous workplace injuries and their development if they occurred. It is important to note that you can simply answer the questions with which you feel comfortable. The purpose of this questionnaire is to help us better understand workplace injury development and find solutions, such as developing a new workplace warm-up and stretching program or implementing new technologies.

#### POTENTIAL RISKS AND DISCOMFORTS

Feelings of anxiety or self-consciousness may occur as a result of having your actions monitored. In the event of discomfort with the use of the heart rate monitor or the watch, accommodations can be made between the researcher and the participant.

Participation in this study is strictly voluntary, meaning you are free to stop being part of the study at any time.

#### POTENTIAL BENEFITS TO SUBJECTS AND/OR SOCIETY

This study aims to understand the physical demands associated with patient handling and other physical tasks performed by caregivers working in long term-care facilities, with the future goal of developing strategies to reduce the high rates of musculoskeletal injury reported among health care providers. The results of this study will make a valuable contribution to current literature, providing a better understanding of the real physical demands of caregivers in a long-term care facility setting. The

database obtained from this study can then be used to develop strategies aimed at reducing the occurrence of work-related musculoskeletal injuries among this working population.

#### CONFIDENTIALITY

Any information that is obtained in connection with this study that can be identified with you will remain completely confidential and will be only disclosed with your permission. Only the investigators will have access to the data. All data will be stored in a locked environment within the Occupational Performance Laboratory in the Faculty of Kinesiology at the Université de Moncton and will remain there for a period of five years, at which point it will be destroyed. A participant pin number will be used in place of your name so that neither you nor your information can be identified. In addition, the results of the study will not include your individual data unless you have given prior consent.

#### PARTICIPATION AND WITHDRAWAL

You can choose whether to be in this study or not. If you volunteer to be in this study, you may withdraw at any time without explanation of why you are withdrawing and without consequences.

This project has been reviewed by the Research Ethics board of the University of New Brunswick and is on file as REB 2024-040 and the Research Ethics board of the Université de Moncton and is on file as REB 2324-070.